CLINICAL TRIAL: NCT02353949
Title: Investigating the Clinical Consequences of Flutemetamol-PET-scanning
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Flutemetamol 2
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease; Dementia
Keywords: Mild cognitive impairment; Alzheimer; PET; Amyloid; Frontotemporal
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flutmetamol Group (Experimental): PET-MR-Scan with 80-140 MBq Flutemetamol before observational period for diagnostic purpose
  Interventions: Drug: Flutemetamol (Vizamyl)

INTERVENTIONS:
Drug: Flutemetamol (Vizamyl) — PET-MR Scan using the radiotracer Flutemetamol (Vizamyl) for diagnostic purpose

SUMMARY:
The study examines subjects where there might be an indication for Amyloid-PET according to the Criteria defined by the Amyloid Imaging Task Force. In these subjects the impact of a Flutemetamol (Vizamyl)-Positron-Emission-Tomography -Scan (PET) on clinical management and disease course will be studied over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Dementia expert considers an Amyloid-scan appropriate according to Amyloid-imaging task force criteria (AIT) after conference with an Amyloid-PET expert
* Preambles of the AIT-Criteria are fulfilled

  1. A cognitive complaint with objectively confirmed impairment
  2. AD as a possible diagnosis, but when the diagnosis is uncertain after a comprehensive evaluation by a dementia expert
  3. When knowledge of the presence or absence of Abeta pathology is expected to increase diagnostic certainty and alter Management

  <!-- -->

  1. Patients with persistent or progressive unexplained MCI
  2. Patients satisfying core clinical criteria for possible AD because of unclear clinical presentation, either an atypical clinical course or an etiologically mixed presentation
  3. Patients with progressive dementia and atypically early age of onset (65 years or less in age)
  4. other situations where preambles of AIT-Criteria are fulfilled
* Diagnosis was established in a memory clinic or by an experienced physician in dementia diagnostics
* The diagnostic procedures comprise in minimum MRI, neuropsychology, routine blood test for exclusion of symptomatic causes
* MMSE >15
* Competency to consent
* Trial partner willing to support study physician
* Written informed consent by both patient and trial partner
* Understanding of German language
* Treating physician willing to collaborate with the study team

Exclusion Criteria:

* Cognitive impairment which can be attributed to another underlying medical condition that renders a possibility of Alzheimer's disease very unlikely (thus violating preamble B)
* Clinically significant Depression (decided upon clinical assessment)
* MRI exclusion criteria
* PET exclusion criteria

  1. Allergy to Flutemetamol or any of the excipients of the solution for injections
  2. History of severe allergic reactions to drugs or allergens
  3. Pregnancy or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Change of ADAS-cog 11 score compared to pre-treatment assessment in Flutemetamol positive subjects with a postscan diagnosis of AD and start of cholinesterase inhibitors as standard treatment. | Three months after initiation of standard treatment

SECONDARY OUTCOMES:
Change of ADCS-ADL score compared to pre-treatment assessment in Flutemetamol positive subjects with a postscan diagnosis of AD and start of cholinesterase inhibitors as standard treatment. | Three months after initiation of standard treatment
Change of ADCS-CGIC score compared to pre-treatment assessment in Flutemetamol positive subjects with a postscan diagnosis of AD and start of cholinesterase inhibitors as standard treatment. | Three months after initiation of standard treatment
Change of MMSE score compared to pre-treatment assessment in Flutemetamol positive subjects with a postscan diagnosis of AD and start of cholinesterase inhibitors as standard treatment. | Three months after initiation of standard treatment

OTHER OUTCOMES:
Comparisons of change from pre-treatment assessment of ADAS-Cog-11 after 6 months in clinical constellations defined by clinical diagnosis and Flutemetamol-status | Six Months after initiation of standard treatment
Comparisons of change from pre-treatment assessment of ADCS-ADL after 6 months in clinical constellations defined by clinical diagnosis and Flutemetamol-status | Six Months after initiation of standard treatment
Comparisons of change from pre-treatment assessment of MMSE after 6 months in clinical constellations defined by clinical diagnosis and Flutemetamol-status | Six Months after initiation of standard treatment
Comparisons of change from pre-treatment assessment of ADCS-CGIC after 6 months in clinical constellations defined by clinical diagnosis and Flutemetamol-status | Six Months after initiation of standard treatment
Change from pre-treatment assessment on the decision regret scale after three months | Three Months after initiation of standard treatment
Change from pre-treatment assessment on the decision regret scale after six months | Six Months after initiation of standard treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hock, MD, Prof., Principal Investigator — University of Zurich, Institute for Regenerative Medicine, Center for Prevention and Dementia Therapy
Locations (1):
- University of Zurich, Institute for Regenerative Medicine, Center for Prevention and Dementia Therapy, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided